CLINICAL TRIAL: NCT00129662
Title: Comprehension and Evaluation of a Pictorial Action Plan for Those With Asthma or Chronic Obstructive Pulmonary Disease
Brief Title: Comprehension and Evaluation of a Pictorial Action Plan for Those With Asthma or COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NHLICX04Q0401103
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Asthma; COPD
Keywords: Pictorial action plan
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Pictorial action plan
  Interventions: Behavioral: Pictorial action plan

INTERVENTIONS:
Behavioral: Pictorial action plan

SUMMARY:
Some five million people in the United Kingdom (U.K.) have asthma. The British Guidelines on Asthma recommend self management education and the issuing of written personal asthma action plans. The use of such self management education has been shown to be associated with an up to 40% reduction in hospitalisation rates and a 20% reduction in Emergency Department attendances and similar benefits in terms of symptoms and time off work. In asthma, the results are best when the patients are provided with a personalised written action plan explaining how to alter their medications according to a variety of circumstances. Chronic obstructive pulmonary disease is a major cause of hospitalisation in the U.K. and is the fourth biggest single cause of death. A recent Cochrane review regarding the value of self management education in COPD has led to equivocal results although it has shown that those with COPD are willing to take control of their own conditions. The reasons for the different outcomes in asthma and COPD may reflect an inadequate number of trials of the wrong type; interventions that were not appropriate or do not work; lack of the use of written action plans; or assessment of benefit using the wrong outcomes.

Given the importance attached to the written action plan, it is essential that such advice is available to all. However, studies of outpatients attending hospitals in the U.K. have shown that 15% may be functionally illiterate and in studies of adults with asthma in the United States (U.S.), 13% have similarly shown to be functionally illiterate. Pictorial advice may therefore be advantageous and, when tested amongst those who are literate, it has been also shown to enhance the recall of spoken medical instructions. The investigators have therefore prepared some pictorial representations which are designed to give advice to those with asthma and COPD about how to recognise the worsening of their conditions and what treatments to alter or initiate as a result. The investigators now need to assess the comprehensibility of those materials amongst a selection of patients with asthma and COPD.

DETAILED DESCRIPTION:
Some five million people in the U.K have asthma. The British Guidelines on Asthma recommend self management education and the issuing of written personal asthma action plans. The use of such self management education has been shown to be associated with an up to 40% reduction in hospitalisation rates and a 20% reduction in Emergency Department attendances and similar benefits in terms of symptoms and time off work. In asthma, the results are best when the patients are provided with a personalised written action plan explaining how to alter their medications according to a variety of circumstances. Chronic obstructive pulmonary disease is a major cause of hospitalisation in the U.K. and is the fourth biggest single cause of death. A recent Cochrane review regarding the value of self management education in COPD has led to equivocal results although it has shown that those with COPD are willing to take control of their own conditions. The reasons for different outcomes in asthma and COPD may reflect an inadequate number of trials of the wrong type; interventions that were not appropriate or do not work; lack of the use of written action plans; or assessment of benefit using the wrong outcomes.

Given the importance attached to the written action plan, it is essential that such advice is available to all. However studies of outpatients attending hospitals in the U.K. have shown that 15% may be functionally illiterate and in studies of adults with asthma in the U.S., 13% have similarly shown to be functionally illiterate. Pictorial advice may therefore be advantageous and when tested amongst those who are literate, it has been also shown to enhance the recall of spoken medical instructions. The investigators have therefore prepared some pictorial representations which are designed to give advice to those with asthma and COPD about how to recognise the worsening of their conditions and what treatments to alter or initiate as a result. The investigators now need to assess the comprehensibility of those materials amongst a selection of patients with asthma and COPD.

Patients will be recruited from two clinics (asthma and COPD) on a Tuesday morning and Thursday afternoon.

On arrival to the Asthma clinic and to the COPD clinic, patients will be given a short information leaflet which they will be invited to read whilst waiting to see the doctor. At the end of the routine consultation they will be asked if they would be willing to help with the study and will be given a patient information sheet and if the patient agrees he/she, will be asked to sign the consent form. The voluntary nature of this and the fact that non-participation will not in any way influence their routine care would be stressed repetitively, both verbally and of course in the patient information leaflet. If the patients were willing to spend a few minutes with the researcher, they would be introduced to the researcher by the consultant in clinic and the interview would either occur on that occasion or at a pre-arranged time to suit the patient. In the first part of the interview, the patient would be given the two pictorial questionnaires to complete which assess the translucency and guessability of the pictogram used for the investigators' pictorial action plans. The second part of the interview would involve explaining to the patient the concept of self management education and personal action plans and a pictorial action plan relevant to the patient would be shown to the patient and he/she would be asked to describe what action should be taken as a result of the pictorial sequences. A series of short questions about the self management plan and his/her preferences for either written or a pictorial plan would be asked. The patient would also be asked to undertake the REALM adult literacy test and demographic data regarding educational attainment, age and ethnicity would also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of spoken English language
* Evidence of respiratory disease (either asthma or COPD)

Exclusion Criteria:

* Poor level of English language; English not first language
* Poor eyesight or literacy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Recall and understanding after pictorial self management education | Baseline only
  information recall after education
Translucency and guessability scores comprehensibility | Baseline
  This outcome measure provides score for each image used in the plan

CONTACTS AND LOCATIONS:
Overall Officials: Martyn R Partridge, MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- NHLI Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roberts NJ, Evans G, Blenkhorn P, Partridge MR. Development of an electronic pictorial asthma action plan and its use in primary care. Patient Educ Couns. 2010 Jul;80(1):141-6. doi: 10.1016/j.pec.2009.09.040. Epub 2009 Oct 29. PMID 19879092